CLINICAL TRIAL: NCT02181322
Title: An Open, Randomised, Four-way Crossover Study in Healthy Volunteers to Evaluate the Effect of Food on the Pharmacokinetics of Meloxicam After a Single p.o. Administration of 22.5 mg Meloxicam Oral Suspension and Dose-proportionality Over a Dosage Range of 7.5 mg to 22.5 mg.
Brief Title: Study to Assess the Effect of Food on the Pharmacokinetics of Meloxicam After Single Administration and to Investigate Dose-proportionality Over a Dosage Range
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.243
Record Dates: First submitted 2014-07-02; First posted 2014-07-03 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

ARMS (4):
- Meloxicam - low dose, fasted (Experimental)
  Interventions: Drug: Meloxicam - low dose
- Meloxicam - medium dose, fasted (Experimental)
  Interventions: Drug: Meloxicam - medium dose
- Meloxicam - high dose, fasted (Experimental)
  Interventions: Drug: Meloxicam - high dose
- Meloxicam - high dose, fed (Experimental)
  Interventions: Drug: Meloxicam - high dose

INTERVENTIONS:
Drug: Meloxicam - low dose
  Arms: Meloxicam - low dose, fasted
Drug: Meloxicam - medium dose
  Arms: Meloxicam - medium dose, fasted
Drug: Meloxicam - high dose
  Arms: Meloxicam - high dose, fasted; Meloxicam - high dose, fed

SUMMARY:
Study to assess the effect of food on the pharmacokinetics of meloxicam after a single p.o. administration of 22.5 mg meloxicam oral suspension and to investigate dose-proportionality over a dosage range of 7.5 mg to 22.5 mg

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Age range from 21 to 50 years
* Broca-Index +- 20%
* In accordance with Good Clinical Practice (GCP) and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Disease of the central nervous system (such a epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial (<= one week prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 mL within four weeks prior to administration or during the trial
* Excessive physical activities (within the last week before study)
* Anl laboratory value outside the reference range of clinical relevance
* History of haemorrhagic diatheses
* History of gastrointestinal ulcer, perforation or bleeding
* History of bronchial asthma

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g sterilisation, intrauterine pessary, oral contraceptives
* Inability to maintain this adequate contraception during the whole study period
* Lactating

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2001-06; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) | up to 96 hours after drug administration
AUC0-infinity (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 96 hours after drug administration
AUC0-tf (Total area under the plasma drug concentration-time curve (AUC) from time of administration (0) to the last quantifiable drug concentration) | up to 96 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 96 hours after drug administration
Terminal rate constant in plasma | up to 96 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 96 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 96 hours after drug administration
MRTtot (Total mean residence time) | up to 96 hours after drug administration
Number of patients with adverse events | up to 10 weeks